CLINICAL TRIAL: NCT01728493
Title: Primary Aldosteronism in General Practice: Organ Damage, Epidemiology and Treatment
Acronym: PAGODE
Status: Completed | Type: Observational
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Principal Investigator, JDeinum, Dr J Deinum, Radboud University Medical Center
Other Study IDs: 40133.091.12
Record Dates: First submitted 2012-11-13; First posted 2012-11-19 (Estimated); Last update posted 2016-04-06 (Estimated); Status verified 2016-04

CONDITIONS: Primary Aldosteronism; Primary Hyperaldosteronism
Keywords: Prevalence; Primary aldosteronism; Organ damage; Mineralocorticoid receptor antagonists
MeSH Terms: conditions — Hyperaldosteronism

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Part 1: - newly diagnosed hypertensive patients in general practice
- Part 2:: * newly diagnosed hypertensive patients with primary aldosteronism
  * newly diagnosed hypertensive patients with essential hypertension
- Part 3:: * newly diagnosed hypertensive patients with normokalemic primary aldosteronism
  * newly diagnosed hypertensive patients with essential hypertension

SUMMARY:
Primary aldosteronism (PA) is the most frequent form of secondary hypertension. It is caused by autonomous secretion of aldosterone, encompassing a group of disorders which is for 99% predominated by unilateral aldosterone-producing adenoma (APA) and bilateral adrenal hyperplasia (BAH). Diagnosis of PA is relevant for two reasons:

1. independent of the level of blood pressure, hypertension due to autonomous aldosterone secretion causes more cardiovascular damage than essential hypertension;
2. PA requires specific treatment: adrenalectomy in case of APA and mineralocorticoid receptor antagonists (MRA) in case of BAH.

Although previously presumed a rare condition (prevalence <1%), PA is now estimated to affect 6 to 20% of the hypertensive population. Given this high prevalence of PA, as well as the amount of cardiovascular damage and the available specific treatment, the question is raised whether screening of PA should be introduced in Dutch general practice. To answer this important question, several issues with regard to PA need to be elucidated:

1. International studies report a prevalence of PA in general practice of 6-13%. Prevalence in the Dutch population is still unknown;
2. Because of underdiagnosis of PA and long delay in diagnosis of PA after recognition of hypertension (mean eight years), data on characteristics of early diagnosed PA are lacking. Proof of early cardiovascular damage would strengthen the case of screening for PA and needs to be studied;
3. Consequently, the diagnostic delay has lead to lack of data on optimal treatment in early PA. In the current guideline (NHG-guideline 'Cardiovascular risk management') a regimen of antihypertensive drugs is advised, and only if hypertension is refractory for >6 months patients are referred. It is unknown if hypertension is resistant to therapy in the initial phase of PA. If not, this would also argue for early biochemical screening for PA, because even if blood pressure is controlled, the detrimental effect of aldosterone itself will go on unopposed. It is therefore required to study the response to antihypertensive drugs (not MRA) in these patients.

DETAILED DESCRIPTION:
Rationale: Primary aldosteronism (PA) is the most frequent form of secondary hypertension. It is caused by autonomous secretion of aldosterone, encompassing a group of disorders which is for more than 99% predominated by unilateral aldosterone-producing adenoma (APA) and bilateral adrenal hyperplasia (BAH). Diagnosis of PA is relevant for two reasons: 1) independent of the level of blood pressure, hypertension due to autonomous aldosterone secretion causes more cardiovascular damage than essential hypertension; 2) PA requires specific treatment: adrenalectomy in case of APA and mineralocorticoid receptor antagonists (MRA) in case of BAH.

Although previously presumed a rare condition (prevalence <1%), PA is now estimated to affect 6 to 20% of the hypertensive population. Given this high prevalence of PA, as well as the amount of cardiovascular damage and the available specific treatment, the question has been raised whether screening of PA should be introduced in Dutch general practice. To answer this important question, several issues with regard to PA need to be elucidated:

1. International studies report a prevalence of PA in general practice of 6-13%. Prevalence in the Dutch population is still unknown;
2. Up to now, the laboratory test for screening for PA, the aldosterone/renin ratio (ARR), is primarily used in secondary care. The relation between the ARR and outcomes in primary care is unknown;
3. Because of underdiagnosis of PA and long delay in diagnosis of PA after recognition of hypertension (mean eight years), data on characteristics of early diagnosed PA are lacking. Indications of early cardiovascular damage would strengthen the case of screening for PA and needs to be studied.

ELIGIBILITY:
Inclusion Criteria:

Part 1:

1. Newly diagnosed hypertensive patients (according to the NHG-guideline 'Cardiovascular risk management');
2. 18 years or older;
3. No use of antihypertensive medication.

Part 2:

1. Patients with increased aldosterone/renin ratio;
2. Positive sodium loading test;
3. Written informed consent.

Part 2 + 3:

1. Patients with normal aldosterone/renin ratio;
2. Normal ARR;
3. Written informed consent.

Part 3:

1. Patients with increased aldosterone/renin ratio;
2. Positive sodium loading test;
3. Normokalemic;
4. Written informed consent.

Exclusion Criteria:

1. Use of antihypertensive medication;
2. Heart failure class II, III or IV (according to the New York Heart Association);
3. Pregnancy or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Newly diagnosed hypertensive patients in general practice (primary care).
Sampling Method: Probability Sample
Enrollment: 700 (Actual)
Dates: Start 2013-09; Primary Completion 2015-12 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
PAGODE part 1: prevalence | 4 months
  Prevalence of primary aldosteronism in newly diagnosed hypertensive patients in Dutch general practice.
PAGODE part 2: organ damage | 4 weeks
  Difference in cardiorenovascular damage in patients with versus without primary aldosteronism, based on a composite of the following parameters:
  1. Left ventricular mass index in g/m2;
  2. Intima-media thickness of carotid artery in mm;
  3. Pulse wave velocity in m/s;
  4. Central aortic blood pressure in mmHg;
  5. Flow-mediated dilation in %;
  6. Albuminuria in mg albumin per mmol creatinin.
PAGODE part 3: blood pressure regulation | 4 months
  Difference in reduction of daytime systolic ambulatory blood pressure measurement (ABPM) in patients with normokalemic primary aldosteronism versus patients with essential hypertension in a standardized treatment regimen during conventional antihypertensive therapy.

SECONDARY OUTCOMES:
PAGODE part 2: organ damage | 4 weeks
  To observe differences between newly diagnosed hypertensive patients with versus without primary aldosteronism in:
  1. Serum potassium;
  2. Low density lipoprotein;
  3. Total cholesterol to high density lipoprotein ratio.
PAGODE part 3: blood pressure regulation | 4 months
  To observe differences between newly diagnosed hypertensive patients with versus without primary aldosteronism in:
  1. Reduction of daytime systolic ABPM in patients with primary aldosteronism versus patients with essential hypertension in a standardized treatment regimen during spironolactone (or eplerenone);
  2. Serum potassium response using conventional antihypertensive medication;
  3. Adverse effects using conventional antihypertensive medication;
  4. Serum potassium response using spironolactone (or eplerenone);
  5. Adverse effects using spironolactone (or eplerenone).

OTHER OUTCOMES:
PAGODE part 2: organ damage | 4 weeks
  To observe differences between newly diagnosed hypertensive patients with versus without primary aldosteronism in:
  1. Serum sodium;
  2. Serum glucose;
  3. Diastolic blood pressure.
PAGODE part 3: blood pressure regulation | 4 months
  To observe differences between newly diagnosed hypertensive patients with versus without primary aldosteronism in:
  1. Reduction in 24 hour ABPM using conventional antihypertensive medication;
  2. Reduction in 24 hour ABPM using mineralocorticoid receptor antagonists.

CONTACTS AND LOCATIONS:
Locations (1):
- Radboud university medical center, Nijmegen, Gelderland, Netherlands